CLINICAL TRIAL: NCT01690442
Title: Couples Based HIV/STI Prevention for Injecting Drug Users in Kazakhstan
Brief Title: HIV Prevention for Injecting Drug Users in Kazakhstan
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Nabila El-Bassel, PhD, Director of the Social Intervention Group, Global Health Research Center of Central Asia, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAD2056
Record Dates: First submitted 2012-09-19; First posted 2012-09-21 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-02

CONDITIONS: HIV; AIDS
Keywords: HIV; AIDS; Prevention
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Couples Based HIV/STI Risk Reduction Intervention (CHSR) (Experimental): The intervention includes a combination of empowerment and couple self-efficacy building strategies, which are employed to help couples overcome resistance to risk reduction.
  Interventions: Behavioral: Couples Based HIV/STI Risk Reduction Intervention (CHSR)
- Renaissance Wellness Promotion (WP) (Active Comparator): This intervention employs a psychoeducational approach to promote wellness, focusing on: maintaining a healthy diet on a low budget, exercising and fitness, stress reducing strategies and specific health related issues that affect IDUs, such as overdose.
  Interventions: Behavioral: Renaissance Wellness Promotion (WP)

INTERVENTIONS:
Behavioral: Couples Based HIV/STI Risk Reduction Intervention (CHSR) — The intervention includes a combination of empowerment and couple self-efficacy building strategies, which are employed to help couples overcome resistance to risk reduction.
  Arms: Couples Based HIV/STI Risk Reduction Intervention (CHSR)
Behavioral: Renaissance Wellness Promotion (WP) — This intervention employs a psychoeducational approach to promote wellness, focusing on: maintaining a healthy diet on a low budget, exercising and fitness, stress reducing strategies and specific health related issues that affect IDUs, such as overdose.
  Arms: Renaissance Wellness Promotion (WP)

SUMMARY:
The proposed study addresses a significant public health threat of HIV, HCV and other STIs among a very high risk population of active IDUs and their sexual partners in Kazakhstan a region that is experiencing one of the fastest rising HIV epidemics in the world. There is a race to develop and implement effective HIV preventive interventions for IDUs and their sexual partners to stem the spread of HIV, HCV and other STIs in Almaty, Shu and other Central Asian towns along drug trafficking routes. The proposed study will test the effectiveness of a couplesbased HIV/STI risk reduction intervention to decrease new cases of HIV and Hepatitis C (HCV) and incidence of sexually transmitted infections (STIs), as well as to reduce unsafe injection practices and increase condom use among injecting drug users (IDUs) and their heterosexual, intimate partners in Kazakhstan.

DETAILED DESCRIPTION:
The proposed study will rigorously test the efficacy of an innovative, couplesbased HIV/STI risk reduction intervention to decrease new cases of HIV and Hepatitis C (HCV) and incidence of sexually transmitted infections (STIs), as well as to reduce unsafe injection practices and increase condom use among injecting drug users (IDUs) and their heterosexual intimate partners in Kazakhstan. Central Asia has experienced one of the fastest growing HIV/AIDS epidemics due to a sharp increase in injection drug use. For the proposed study, the participants will be 400 IDUs and their heterosexual intimate partners. These 400 couples will be randomized to one of two interventions: a 5session couplesbased HIV/STI risk reduction intervention or a 5session couplesbased wellness promotion intervention, which will serve as a control condition. Participants will be assessed with repeated measures at baseline, 3, 6, and 12months postintervention. The primary behavioral outcomes are selfreported proportion of injection acts in which needles or syringes are shared in the past 90 days and proportion of condom protected acts of sexual intercourse in the past 90 days. The primary biological outcomes are the rate of new HIV and HCV cases, and the cumulative incidence of Chlamydia, gonorrhea, and syphilis over the 12month postintervention period. The proposed study will advance the understanding of HIV/HCV/STI risk reduction among IDUs and thereby may help to stem the rising epidemic of HIV, HCV, and STIs in Kazakhstan and Central Asia.

ELIGIBILITY:
Inclusion Criteria:

* Couples are eligible to participate if both partners are aged 18 or older
* both partners identify each other as their main partner of the opposite sex and someone whom the participant considers a boy/girlfriend, spouse, lover and/ or parent of his/her child
* the relationship has existed at least 3 months
* each partner intends to remain together for at least 12 months
* at least one partner reports having had unprotected vaginal or anal intercourse with the other partner at least once in the previous 90 days
* at least one partner reports injecting drugs in the past 90 days
* neither partner has plans to relocate beyond a reasonable distance from the study site

Exclusion Criteria:

* Couples are excluded if either partner shows evidence of significant psychiatric, physical or neurological impairment that would limit effective participation as confirmed on a MiniMental State Examination and/or Quick Test
* either partner reports severe physical violence perpetrated by the other partner in the past year on the Revised Conflict Tactics Scale
* either partner is unable to commit to participate in the study through to completion
* either partner reports that the couple is planning a pregnancy within the next 18 months
* either partner is not fluent in Russian as determined during Informed Consent
* both partners do not meet all eligibility criteria or meet one or more exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2008-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
The proportion of condom protected acts of vaginal and anal intercourse | 12 months
The number of incidents of unclean syringes or needles in the past 90 days | 12 months
Proportion of injection acts in which unclean needles or syringes were used in the past 90 days | 12 months
The number of acts of unprotected vaginal and anal intercourse during the 90 days prior to the assessment period | 12 months

SECONDARY OUTCOMES:
Number of people participants shared needles or syringes with in the past 90 days | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Nabila El-Bassel, Principal Investigator — Columbia University
Locations (1):
- Global Health Research Center of Central Asia, Almaty, Kazakhstan